CLINICAL TRIAL: NCT00103753
Title: A Randomized, Placebo Controlled, Double Blind Trial of the Effect of Combined Therapy With Deferoxamine and Deferiprone on Myocardial Iron in Thalassemia Major Using Cardiovascular Magnetic Resonance
Brief Title: Combined Chelation Treatment With Deferiprone and Deferoxamine in Thalassemia Major
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: CORDA, The Heart Charity (Other); The Cooley's Anemia Foundation, (Other); Apotex Inc. (Industry); The UK Thalassemia Society (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 02 065
Record Dates: First submitted 2005-02-14; First posted 2005-02-15 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-02

CONDITIONS: Beta-Thalassemia
Keywords: Randomized Controlled Trial; Deferiprone; Deferoxamine; Iron chelation; Beta Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia | interventions — Deferiprone

INTERVENTIONS:
Drug: deferiprone

SUMMARY:
Thalassemia major is a genetic disorder affecting hemoglobin synthesis, rendering individuals dependent upon lifelong blood transfusions. Consequently, iron overload occurs and patients have shortened life expectancy with the most common cause of death being heart failure. This trial tests whether the combination of traditional therapy (deferoxamine) with a newer drug (deferiprone) will prove more effective in removing cardiac iron than deferoxamine alone.

DETAILED DESCRIPTION:
Thalassemia Major (TM) is a hereditary anemia resulting from a single gene defect that results in abnormal red cell production. The survival of affected individuals is dependent upon lifelong blood transfusions. Unfortunately, this causes total body iron overload, and 50% of the patients in the UK are dead by the age of 35. Approximately 70% of these deaths result from heart failure which results as a consequence of cardiac iron toxicity.

A Cardiovascular Magnetic Resonance (CMR) technique (which exploits the fact that T2* signal decay relates to tissue iron) developed at the Royal Brompton Hospital provides a non-invasive and reproducible assessment of cardiac iron. CMR therefore provides a very useful method to assess response to new treatments in this condition. Using cardiac T2* as a primary endpoint, we will investigate whether the oral chelator, deferiprone in combination with traditional treatment (deferoxamine), is superior in removing cardiac iron as compared to deferoxamine alone. This trial will provide the first randomized controlled, double-blinded, evidence for the efficacy of combination treatment in TM.

ELIGIBILITY:
Inclusion Criteria:

* Beta thalassemia major
* Maintaining pre-transfusion hemoglobin of 9 g/dL
* Myocardial T2* between 8 and 20 ms
* Ability to give informed consent
* Male or female
* Age >18 years
* Any ejection fraction
* Confirmation of effective contraception throughout the trial (both men and women)

Exclusion Criteria:

* Implant incompatible with MR (magnetic resonance), such as pacemaker, claustrophobia, or other condition making CMR impossible or inadvisable
* Neutropenia within 12 months (ANC <1.5 x10^9/L), unless normal at screening
* Thrombocytopenia within 12 months (<50 x10^9/L), unless normal at screening
* Liver enzymes > 3 times upper limit of normal
* Patients who have previously received deferiprone for a total of more than 6 months over the last 5 years.
* Patients with a previous reaction to deferiprone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65
Dates: Start 2004-05; Study Completion 2005-06

PRIMARY OUTCOMES:
Myocardial T2*

SECONDARY OUTCOMES:
Liver T2*
LV and RV volumes and function in systole and diastole
Brachial artery reactivity
B-type natriuretic peptide
Patient compliance
Adverse events
Success of blinding

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Microcitemico, Via Jenner, Cagliari, Sardinia, Italy

REFERENCES:
- [Derived] Tanner MA, Galanello R, Dessi C, Smith GC, Westwood MA, Agus A, Pibiri M, Nair SV, Walker JM, Pennell DJ. Combined chelation therapy in thalassemia major for the treatment of severe myocardial siderosis with left ventricular dysfunction. J Cardiovasc Magn Reson. 2008 Feb 25;10(1):12. doi: 10.1186/1532-429X-10-12. PMID 18298856